CLINICAL TRIAL: NCT07341633
Title: Efficacy of Artificial Intelligence-Based Digital Therapeutics Versus Traditional Schroth Exercises for Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial
Brief Title: AI-Based Digital Therapeutics vs. Traditional Schroth Exercises for Adolescent Idiopathic Scoliosis
Acronym: AIS-DTx-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Ma Ruisi, Lecturer, Jinan University Guangzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GWCMC-2025-497A01
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Digital Therapeutics; Artificial Intelligence; Schroth Method; Tele-rehabilitation; Computer Vision; Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: A parallel-group, single-blind randomized controlled trial comparing an AI-based digital therapeutic intervention against a standard care control group.
Who Masked: Outcomes Assessor
Masking Description: Due to the visible nature of the exercise intervention, it is not possible to blind participants or care providers. To minimize detection bias, the primary outcome (Cobb angle) will be assessed by independent radiologists who are strictly blinded to group allocation and the timing of the radiographs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Outpatient Schroth Therapy (Active Comparator): Participants receive standard conservative care based on Schroth Best Practice guidelines. This involves an initial 60-minute comprehensive evaluation, followed by a personalized home exercise program (30 minutes daily). Participants attend monthly supervised sessions at the outpatient clinic for manual prescription adjustments by a certified therapist .
  Interventions: Procedure: Standard Outpatient Schroth Therapy
- AI-Based Digital Therapeutics (AI-DTx) (Experimental): Participants utilize a smartphone application to capture standardized photos every two weeks. An AI algorithm (MediaPipe-based) processes these images to classify curve patterns and assign personalized exercise modules. The system uses a "Human-in-the-Loop" workflow where a Clinical Research Assistant verifies the AI-generated prescription before release. Dosing intensity is adaptively adjusted based on metric changes.
  Interventions: Device: AI-Based Digital Therapeutic System

INTERVENTIONS:
Device: AI-Based Digital Therapeutic System — A smartphone-based digital therapeutic application that utilizes computer vision (MediaPipe Framework) to capture and analyze patient posture bi-weekly. The system employs a hierarchical triage logic to classify curve patterns and assign personalized Schroth-based exercise modules. It features a "Human-in-the-Loop" safety protocol where a Clinical Research Assistant validates the AI-generated prescription before release. The exercise dosing (intensity and props) is adaptively adjusted based on the calculated metric changes (NSI) every two weeks .
  Arms: AI-Based Digital Therapeutics (AI-DTx)
Procedure: Standard Outpatient Schroth Therapy — Standard conservative management based on the SOSORT and Schroth Best Practice guidelines. Participants undergo an initial 60-minute comprehensive evaluation and education session. The intervention consists of a daily home exercise program (30 minutes/day) and mandatory monthly face-to-face supervised sessions at the outpatient clinic, where a certified therapist manually adjusts the exercise prescription based on clinical progression .
  Arms: Standard Outpatient Schroth Therapy

SUMMARY:
This randomized controlled trial (RCT) evaluates the efficacy of a novel Artificial Intelligence (AI)-based digital therapeutic system compared to traditional outpatient Schroth exercises for the treatment of Adolescent Idiopathic Scoliosis (AIS). The intervention utilizes a smartphone application with computer vision technology to perform remote, personalized posture analysis and generate adaptive exercise prescriptions. The study aims to determine if this "Human-in-the-Loop" AI model demonstrates superior clinical outcomes in controlling spinal curve progression and improving treatment adherence compared to standard conservative care over a 6-month period.

DETAILED DESCRIPTION:
Background: Adolescent Idiopathic Scoliosis (AIS) requires long-term conservative management to prevent curve progression. While Physiotherapeutic Scoliosis Specific Exercises (PSSE), such as the Schroth method, are the gold standard, their efficacy is often limited by accessibility barriers and suboptimal adherence.

Study Design: This is a parallel-group, single-blind randomized controlled trial. A total of 300 eligible adolescents (aged 10-18, Cobb angle 10-30°, Risser sign 0-2) will be randomized in a 1:1 ratio into an Intervention Group or a Control Group.

Interventions:

Intervention Group (AI-DTx): Participants utilize a smartphone application to capture standardized photos every two weeks. An AI algorithm (based on MediaPipe) extracts skeletal landmarks to classify curve patterns and assign personalized exercise modules. The system features a "Check-and-Adjust" matrix to adapt exercise intensity based on metric changes. A Clinical Research Assistant (Human-in-the-Loop) verifies all prescriptions for safety before release.

Control Group (Standard Care): Participants receive standard outpatient Schroth therapy, involving daily home exercises and monthly supervised clinic visits, following SOSORT guidelines.

Objectives: The primary objective is to evaluate the absolute change in the major curve Cobb angle from baseline to six months. Secondary outcomes include the Angle of Trunk Rotation (ATR), trunk appearance perception (TAPS), quality of life (SRS-22r), and adherence rates. The study hypothesizes that the AI-driven intervention will demonstrate superior efficacy and adherence compared to traditional outpatient care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Adolescent Idiopathic Scoliosis (AIS).
2. Age between 10 and 18 years (inclusive).
3. Cobb angle of the major curve between 10° and 30°.
4. Risser sign 0-2 (indicating skeletal immaturity).
5. Ability to operate a smartphone and follow instructions for the digital therapeutic application.
6. Patient and legal guardian provide written informed consent.

Exclusion Criteria:

1. Non-idiopathic scoliosis (e.g., congenital, neuromuscular, or syndromic etiology).
2. History of prior spinal surgery or currently scheduled for surgery.
3. Contraindications to exercise therapy (e.g., cardiac or respiratory insufficiency).
4. Severe cognitive or psychiatric disorders that prevent compliance with the protocol.
5. Currently receiving other scoliosis-specific treatments (e.g., bracing) outside of the study protocol (unless stratified).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Absolute Change in Major Curve Cobb Angle | 0,3,5,6month
  Measured on standardized standing posteroanterior full-spine radiographs. The Cobb angle is the angle formed between the upper endplate of the most tilted upper vertebra and the lower endplate of the most tilted lower vertebra. Measurements are performed in degrees by independent radiologists who are blinded to group allocation. A negative value indicates a reduction (improvement) in the spinal curve.

SECONDARY OUTCOMES:
Treatment Adherence Rate | 0,3,5,6 months
  Calculated as the percentage of completed exercise sessions relative to the prescribed sessions. For the Intervention group, adherence is logged automatically by the app via computer vision verification. For the Control group, adherence is self-reported via paper logs.
Change in Angle of Trunk Rotation (ATR) | 0,3,5,6 months
  Measured using a Scoliometer during the Adam's Forward Bend Test. The maximum rotation angle of the trunk is recorded in degrees.
Change in Quality of Life (SRS-22r Score) | 0,3,5,6 months
  Assessed using the Scoliosis Research Society-22 revised (SRS-22r) questionnaire. The score ranges from 1 to 5, with higher scores indicating better patient outcomes across domains of function, pain, self-image, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Shu, MD, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided